CLINICAL TRIAL: NCT04349618
Title: Open Label Randomized Controlled Trial of Ultraprotective Ventilation Without Extracorporeal Circulation in Patients With COVID 19 Pneumonia and Moderate to Severe ARDS
Brief Title: Ultraprotective Ventilation Without Extracorporeal Circulation During COVID 19 Pneumonia
Acronym: VT4COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL20_0322
Record Dates: First submitted 2020-04-08; First posted 2020-04-16 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome; COVID19; Sars-CoV2; Pneumonia
Keywords: COVID19; ARDS; MECHANICAL VENTILATION; ULTRAPROTECTIVE VENTILATION
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19; Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROTECTIVE VENTILATION (Active Comparator): Protective ventilation with tidal volume 6 mL/kg of predicted body weight
  Interventions: Other: PROTECTIVE VENTILATION
- ULTRAPROTECTIVE VENTILATION (Experimental): Ultraprotective ventilation with tidal volume reduction down to 4 mL/kg further adjusted to keep plateau pressure below 30 cm H2O and pH above 7.20
  Interventions: Other: ULTRAPROTECTIVE VENTILATION

INTERVENTIONS:
Other: PROTECTIVE VENTILATION — Protective ventilation with tidal volume 6 mL/kg of predicted body weight further adjusted to keep plateau pressure below 30 cm H2O and pH above 7.20, and PEEP set using the PEEP FiO2 table of the ARMA trial
  Arms: PROTECTIVE VENTILATION
Other: ULTRAPROTECTIVE VENTILATION — Ultraprotective ventilation with tidal volume reduction down to 4 mL/kg further adjusted to keep plateau pressure below 30 cm H2O and pH above 7.20, and PEEP set using the PEEP FiO2 table of the ARMA trial
  Arms: ULTRAPROTECTIVE VENTILATION

SUMMARY:
Mortality of COVID-19 pneumonia with acute respiratory distress syndrome (ARDS) is extremely high in preliminary reports amounting to 50-60%. Duration of mechanical ventilation in these patients appears to exceed standard duration of mechanical ventilation in non-COVID-19 ARDS patients, suggesting that COVID-19 patients may be particularly at risk for ventilator-induced lung injury. Treatment of COVID-19 ARDS patients is to date mainly supportive with protective mechanical ventilation (ventilation with low tidal volume (VT) i.e. 6 ml/kg of predicted body weight (PBW) and plateau pressure control below 30 cm H2O).

Mechanical ventilation with VT reduction below 6 ml/kg PBW in ARDS may reduce alveolar strain, driving pressure and hence ventilator-induced lung injury. Investigators recently performed a multicenter pilot study on 34 moderately severe to severe ARDS patients. This study demonstrated that ultraprotective ventilation with ultra-low VT (≤4.2 ml/kg PBW) without extracorporeal circulation may be applied in approximately 2/3 of the patients, with a 4 cmH2O median reduction in driving pressure, at the price of transient episodes of severe acidosis in approximately 1/3 of the patients. Investigators hypothesized that ultraprotective ventilation without extracorporeal circulation may reduce the mortality at day-90 and increase the number of days free from mechanical ventilation (VFD) at day-60, as compared to protective ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* ARDS according to the Berlin definition
* COVID-19 pneumonia confirmed by RT-PCR
* Acute respiratory failure not fully explained by left ventricular failure or sodium overload
* Bilateral pulmonary radiological opacities not fully explained by pleural effusions or atelectasis or nodules
* Invasive mechanical ventilation with PaO2/FiO2 ≤ 150 mm Hg and PEEP ≥ 5 cm H2O with a tidal volume below or equal to 6 ml per kilogram of predicted body weight
* Continuous intravenous sedation as part of ARDS treatment

Exclusion Criteria:

* Exclusion criteria related to ARDS history

  * ARDS onset more than 48 hours before inclusion
  * previous inclusion in present study
* Exclusion criteria related to ARDS severity or complications

  * arterial pH < 7.21 despite respiratory rate set to 35/min at the time of inclusion
  * patient under any extracorporeal CO2 removal technique or ECMO
  * pneumothorax or bronchopleural fistula
* Exclusion criteria related to comorbidities

  * suspected intracranial hypertension
  * severe chronic obstructive pulmonary disease defined by a GOLD score ≥ 3
  * chronic respiratory failure under home oxygen or non-invasive ventilation
  * chronic respiratory failure requiring long term oxygen or non-invasive ventilation
  * obesity with body weight over height ratio greater than 1 kg/cm
  * sickle cell disease
  * bone marrow transplant < 6 months
  * burn injury with extension greater than 30% of body surface area
  * cirrhosis with Child-Pugh score C
  * advance directives to withhold or withdraw life sustaining treatment
* Exclusion criteria related to legislation

  * Patient under an exclusion period relative to participation to another clinical trial, or inclusion into a clinical trial interfering with the ventilatory strategies
  * pregnancy, lactating women
  * patient under a legal protective measure.
  * lack of affiliation to social security as required by French regulation
  * lack of written informed consent by patient or next of kin (unless if recourse to the emergency procedure in the absence of a loved one)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
A composite score based on all-cause mortality and the number of ventilator free-days (VFD) | Day 90
  For an alive patient at day 90, the score will be built as follow: a value +1 will be given for comparisons to dead patients and alive patients with a lower number of VFD. For comparisons to alive patients with a higher number of VFD a value -1 will be given and in case of identical number of VFD a value 0 will be given. For a dead patient a value -1 will be given for comparisons to alive patients and 0 for comparisons to dead patients. For a given patients the score will correspond to the sum of values resulting to the comparison to all patients of the other group. A higher score indicates a more favorable result.

SECONDARY OUTCOMES:
All-cause mortality (intention to treat) | 90-day after inclusion
  All-cause mortality with analysis in intention to treat, i.e. each patient will be analyzed in his initial randomization group regardless of whether the allocated strategy was effectively applied or not.
Ventilator-free days (VFD) | day 60 after inclusion
  VFD will be computed as follows from the day of inclusion:
  VFD= 0 if the patient dies between inclusion and day 60 VFD = 60-x if the patient is successfully weaned from invasive mechanical ventilation x days after inclusion. Successful weaning from mechanical ventilation is defined by extubation without reintubation within at least 48 hours (or weaning from mechanical ventilation for at least 48 hours in patients with tracheostomy) VFD= 0 if the patient is mechanically ventilated for more than 60 days after inclusion
All-cause mortality with per protocol analysis | 90-day
  Per protocol analysis will be carried out by comparing the group of patients in whom median daily tidal volume from inclusion to weaning of deep sedation will be lower of equal to 4.2 ml/kg of predicted body weight to the group of patients in whom median tidal volume from inclusion to weaning of deep sedation will be greater than 4.2 ml/kg of predicted body weight, whatever the patients' initial randomization group.
  Weaning of deep sedation is defined by a Richmond Agitation Sedation (RASS) score greater than -3 for at least 48 hours.
Time to successful extubation | 60 days
  Successful extubation is defined by extubation without reintubation within at least 48 hours (or weaning from mechanical ventilation for at least 48 hours in patients with tracheostomy) Data will be right censored at 60 days and death will be taken into account as a competing risk.
Length of hospital stay | 90 days
  Data will be right censored at 90 days and death will be taken into account as a competing risk.
Respiratory parameters assessed daily from inclusion to weaning of deep sedation or 14 days whichever comes first | 14 days
  Weaning of deep sedation is defined by a Richmond Agitation Sedation (RASS) score greater than -3 for at least 48 hours.
Daily sedation dose during the first 14 days of the study | 14 days
  Doses of the following drugs used for deep sedation will be assessed daily: midazolam, propofol and opioid. Opioid dose will be expressed as morphine equivalent with the following conversion factor: 1µg of sufentanil = 10 µg of fentanyl = 1 mg of morphine
Rate of use of rescue therapies | 14 days
  Rescue therapies are any therapy among the following ones: neuromuscular blocking agents, prone position, nitric oxide, recruitment maneuvers, ECMO
Incidence density rate of severe mixed acidosis | ICU stay
  Severe mixed acidosis is defined by the association of pH<7.15 and PaCO2>45 mm Hg.
Incidence density rate of ventilator associated pneumonia | ICU stay
  Ventilator associated pneumonia will be defined as any pneumonia acquired under mechanical ventilation after inclusion.
Incidence density rate of acute cor pulmonale | ICU stay
  Acute cor pulmonale is defined by the association of right ventricle dilatation (right ventricle surface / left ventricle surface >0,6) and septal dyskinesia assessed by echocardiography
Incidence density rate of barotrauma | ICU stay
  Barotrauma is defined by any pneumothorax OR pneumomediastinum OR subcutaneous emphysema, OR pneumatocele of more than 2 cm detected on image examinations.
Incidence density rate of any serious adverse events | ICU stay
  Serious adverse event is any life threatening event OR any event resulting in death.
Cognitive impairment assessed by phone call using the Telephone Montreal Cognitive Assessment (T-MoCA) test | Day 365 after inclusion
  The Telephone Montreal Cognitive Assessment score will be assessed by phone call. The total score ranges from 0 to 30; higher scores being associated to a better outcome.
Quality of life assessed by the RAND 36-Item Health Survey (SF-36) score | Day 365 after inclusion
  The RAND 36-Item Health Survey (SF-36) score will be assessed by phone call. The score ranges from 0 to 100; higher scores being associated to a better outcome.
Post-traumatic stress disorder assessed by the Impact of Event Scale - revised (IES-R) score by phone call | Day 365 after inclusion
  The Impact of Event Scale - revised (IES-R) score will be assessed by phone call. The total score ranges from 0 to 88; higher scores being associated to a worse outcome.
Cost-efficacy ratio of the innovative strategy compared to the reference strategy | Day 90 after inclusion
  The cost-efficacy ratio will be computed as the ratio of cost difference on efficacy difference between the intervention arm and the reference arm. The costs taken into account will be the direct hospitalized costs. The efficacy will be assessed as the number of days alive free from mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Service de Médecine Intensive Réanimation CHU Gabriel Montpied, Clermont-Ferrand
  - Service de Médecine Intensive Réanimation Hôpital Michallon - CHU Grenoble Alpes, La Tronche
  - Service de Médecine Intensive Réanimation Hôpital Edouard Herriot Hospices Civils de Lyon, Lyon
  - Service de Réanimation Chirurgicale Hôpital Edouard Herriot Hospices Civils de Lyon, Lyon
  - Service de Médecine Intensive Réanimation Hôpital de la Croix Rousse Hospices Civils de Lyon, Lyon
  - Service de Réanimation Chirurgicale Hôpital de la Croix Rousse Hospices Civils de Lyon, Lyon
  - Service de réanimation Polyvalente Centre Hospitalier Saint Joseph-Saint Luc, Lyon
  - Service de Réanimation Clinique de la Sauvegarde, Lyon
  - Service de Réanimation Polyvalente Centre Hospitalier Lyon Sud Hospices Civils de Lyon, Pierre-Bénite
  - Service de Réanimation Centre hospitalier Annecy Genevois, Pringy
  - Service de Médecine Intensive Réanimation Hôpital Nord - CHU Saint-Etienne, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Richard JC, Terzi N, Yonis H, Chorfa F, Wallet F, Dupuis C, Argaud L, Delannoy B, Thiery G, Pommier C, Abraham P, Muller M, Sigaud F, Rigault G, Joffredo E, Mezidi M, Souweine B, Baboi L, Serrier H, Rabilloud M, Bitker L; VT4COVID collaborators. Ultra-low tidal volume ventilation for COVID-19-related ARDS in France (VT4COVID): a multicentre, open-label, parallel-group, randomised trial. Lancet Respir Med. 2023 Nov;11(11):991-1002. doi: 10.1016/S2213-2600(23)00221-7. Epub 2023 Jul 12. PMID 37453445
- [Derived] Richard JC, Yonis H, Bitker L, Roche S, Wallet F, Dupuis C, Serrier H, Argaud L, Thiery G, Delannoy B, Pommier C, Abraham P, Muller M, Aubrun F, Sigaud F, Rigault G, Joffredo E, Mezidi M, Terzi N, Rabilloud M. Open-label randomized controlled trial of ultra-low tidal ventilation without extracorporeal circulation in patients with COVID-19 pneumonia and moderate to severe ARDS: study protocol for the VT4COVID trial. Trials. 2021 Oct 11;22(1):692. doi: 10.1186/s13063-021-05665-z. PMID 34635128